CLINICAL TRIAL: NCT00902603
Title: Registry to Prospectively Evaluate Use of Ventavis® in Patients With Pulmonary Arterial Hypertension
Brief Title: Ventavis® Registry Protocol
Acronym: RESPIRE
Status: Terminated | Type: Observational
Why Stopped: low enrollment and difficulty recruiting eligible patients in adequate time
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-063A501
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; Ventavis®; iloprost
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with WHO Group I pulmonary arterial hypertension (PAH) who have been receiving therapy with Ventavis® for at least 3 months.
  Interventions: Drug: Commercial Ventavis® (iloprost)

INTERVENTIONS:
Drug: Commercial Ventavis® (iloprost) — Commercial Ventavis® (iloprost) administered via portable nebulizer (I-neb® AAD® system using the power disc-6)

SUMMARY:
The Ventavis® (iloprost) Registry is a multicenter, observational, U.S.-based study that longitudinally follows patients with pulmonary arterial hypertension (PAH) who have been receiving therapy with Ventavis® for at least 3 months. Patients diagnosed with WHO Group I PAH who are on a stable regimen of commercial Ventavis® will be followed for a maximum of 2 years from the time of enrollment. Data will be collected via patient interview and review of the medical record. Quarterly data collection will include capture of medications and Ventavis® adherence data.

DETAILED DESCRIPTION:
The Ventavis® (iloprost) Registry is a multicenter, observational, U.S.-based study that longitudinally follows patients with pulmonary arterial hypertension (PAH) who have been receiving therapy with Ventavis® for at least 3 months. Patients diagnosed with WHO Group I PAH and who are on a stable regimen of commercial Ventavis® will be followed for a maximum of 2 years from the time of enrollment. All data will be collected via patient interview and/or review of the medical record, as well as from I-neb® downloads using INSIGHT software. Adherence with Ventavis® will be compared before and after targeted instruction on inhalation techniques by a respiratory therapist or designee, as well as before and after participation in PAH patient support groups (if applicable). Quarterly data collection will include capture of PAH and non-PAH medications and Ventavis® adherence data; Ventavis® adherence data will also be collected one month after study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Have a current diagnosis of WHO Group I PAH
2. Have initiated therapy with commercial Ventavis® administered via portable nebulizer at least 3 months prior to study enrollment, either with commercial product or from participation in Actelion's Clinical Study AC-063A302
3. Age > or = 18 years old at the time of enrollment

Exclusion Criteria:

1. Meet the criteria for inclusion into WHO Groups II, III, IV or V PAH
2. Are not currently on commercial Ventavis®
3. Have initiated therapy with commercial Ventavis® administered via portable nebulizer less than 3 months prior to study enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2009-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Adherence with instructions for use of Ventavis® | 2 years

SECONDARY OUTCOMES:
Persistence of use of Ventavis® | 2 years